CLINICAL TRIAL: NCT02337803
Title: Band Together: Randomized Control Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A similar study was funded by PCORI so PI decided to not begin this study.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine and Public Health Sciences; Division Chief of General Internal Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB1056
Record Dates: First submitted 2015-01-08; First posted 2015-01-14 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Age 65 and Older; Strength Training
Keywords: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength Training Group (Experimental): Participants will meet three times a week for one hour strength training sessions for twelve weeks.
  Interventions: Behavioral: Strength Training Program; Behavioral: Usual Care
- Usual Care (Active Comparator): Participants will be given access to the strength training program after the twelve week study ends.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Strength Training Program — The strength training program consists of 6 exercises using resistance bands three times a week
  Arms: Strength Training Group
Behavioral: Usual Care — Will continue daily physical activity and complete surveys online

SUMMARY:
The study will aim to determine the effectiveness of a strength training program using resistance bands to increase strength in adults ≥65 years old

DETAILED DESCRIPTION:
Older adults in the US are in a difficult situation that is historically unprecedented. People born in 1930 were expected to live to age 59, yet they will live to an average age of 79. These dramatic survival increases, due to immunizations, antibiotics and other innovations [Centers for Disease, 2011], have occurred at the same time as dramatic reductions in daily energy expenditures, due to automobiles, washing machines and other labor-saving devices [Archer, 2013]. This has left adults living longer, yet weaker, less fit and more obese. In fact, most residents of nursing homes are not there because of dementia. Only 40% of long-term care facility residents in 2010 were diagnosed with dementia [Caffrey, 2012] and many of whom had a level of dementia which would not require nursing home placement by itself. Most residents of long-term care facilities, rather, are there because they lack the strength and fitness to care for themselves. As baby boomers retire, these factors are anticipated to greatly increase the need for long-term care, highlighted in a report from a Deloitte Consulting in 2010: "Medicaid Long-term Care: The ticking time bomb" [Keckley, 2010]. This pilot study will measure a significant increase in strength with the use of a 12 week strength training program.

ELIGIBILITY:
Inclusion Criteria:

* Fluently read and speak English
* Willing to drive 3 times a week to Hershey Medical Center for most weeks
* Have a primary care physician
* Currently exercise ≤60 min per week

Exclusion Criteria:

* Doctor has said you have a heart condition and should only do physical activity recommended by doctor
* Feel pain in chest when doing physical activity
* Unable to obtain doctor's consent
* Currently participating in an exercise program
* Plans to move in the next 6 months
* Weight > 250
* Currently exercise ≥60 min per week

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
One Repetition Maximum | 12 weeks

SECONDARY OUTCOMES:
Bow and Arrow Strength Test | 12 weeks
Hand Grip Test | 12 weeks

OTHER OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) | 12 weeks
  survey
National Health Interview Surveys | 12 weeks
  survey
Physical Activity Scale for the Elderly (PASE) | 12 weeks
  survey
Cognitive Impairment Questionnaire | 12 weeks
  survey

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Hershey Medical Center, Hershey, Pennsylvania, United States